CLINICAL TRIAL: NCT00911677
Title: Does Apolipoprotein E Genotype Predict Delirium and Postoperative Cognitive Dysfunction?
Brief Title: Does APOE-e4 Predict Delirium and Cognitive Dysfunction After Surgery?
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); University of Ottawa (Other)
Responsible Party: Gregory L Bryson, Department of Anesthesiology, The Ottawa Hospital
Other Study IDs: OHREB 2004800-01H
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction
Keywords: Delirium (MeSH Unique ID D003693); Cognition Disorders (MeSH Unique ID D003072); Postoperative Complications (MeSH Unique ID D011183); Apolipoproteins E (MeSH Unique ID D001057)
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications; Cognition Disorders; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open Aortic Repair: Patients 60 years of age and older undergoing open repair of the abdominal aorta

SUMMARY:
Patients with the APOE-ε4 genotype are at increased risk of both vascular dementia and peripheral vascular disease. Patients undergoing major vascular surgery are at particularly high risk of delirium and other, more subtle, changes in cognitive function following surgery. The hypothesis of this trial is that the APOE-ε4 genotype is associated with both delirium and postoperative cognitive dysfunction (POCD).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or greater
* Open repair of the abdominal aorta

Exclusion Criteria:

* refusal;
* planned endovascular repair;
* emergency surgery;
* previous diagnosis of dementia, Parkinson's disease, or psychiatric illness;
* active alcohol or substance abuse; and
* physical inability to complete neuropsychometric testing.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 60 years of age or greater undergoing open repair of the abdominal aorta at an academic tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Delirium as assessed by the Confusion Assessment Method | 7 days postoperatively

SECONDARY OUTCOMES:
POCD as assessed by a battery of 9 neuropsychometric tests | 7 days postoperatively
POCD as assessed by a battery of 9 neuropsychometric tests | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Bryson, MD, FRCPC, Principal Investigator — Department of Anesthesiology, The Ottawa Hospital
Locations (1):
- The Ottawa Hospital - Civic Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Bryson GL, Wyand A, Wozny D, Rees L, Taljaard M, Nathan H. A prospective cohort study evaluating associations among delirium, postoperative cognitive dysfunction, and apolipoprotein E genotype following open aortic repair. Can J Anaesth. 2011 Mar;58(3):246-55. doi: 10.1007/s12630-010-9446-6. Epub 2011 Jan 11. PMID 21222188
- [Derived] Bryson GL, Wyand A, Wozny D, Rees L, Taljaard M, Nathan H. The clock drawing test is a poor screening tool for postoperative delirium and cognitive dysfunction after aortic repair. Can J Anaesth. 2011 Mar;58(3):267-74. doi: 10.1007/s12630-010-9448-4. Epub 2010 Dec 31. PMID 21194015